CLINICAL TRIAL: NCT03135652
Title: Consolidative Radiotherapy for Colorectal Cancer Liver Metastases Receiving Surgery or Radiofrequency Ablation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate patient enrollment
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of Gastrointestinal Oncology Department, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRLM-AR1
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Radiotherapy; Colorectal Cancer; Liver Metastases
Keywords: Radiotherapy; Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiotherapy; Drug Therapy; Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: adjuvant radiotherapy:SBRT chemotherapy:mFolfox6/ CAPEOX/ Folfiri±cetuximab or bevacizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemoradiotherapy (Experimental): radiotherapy: adjuvant SBRT of liver lesions; chemotherapy: mFolfox6/ CAPEOX/ Folfiri±cetuximab or bevacizumab, 2 months for neoadjuvant treatment and 4 months for adjuvant treatment
  Interventions: Radiation: adjuvant SBRT; Drug: Chemotherapy
- chemotherapy (Active Comparator): chemotherapy: mFolfox6/ CAPEOX/ Folfiri±cetuximab or bevacizumab, 2 months for neoadjuvant treatment and 4 months for adjuvant treatment
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Radiation: adjuvant SBRT — adjuvant SBRT of liver lesions
  Other Names: radiotherapy
  Arms: chemoradiotherapy
Drug: Chemotherapy — mFolfox6/ CAPEOX/ Folfiri±cetuximab or bevacizumab, 2 months for neoadjuvant treatment and 4 months for adjuvant treatment
  Other Names: neoadjuvant chemotherapy and adjuvant chemotherapy

SUMMARY:
This study is a randomized phase II trial to evaluate the efficacy of adjuvant consolidative radiotherapy in colorectal cancer liver metastasis (CRLM) patients after chemotherapy combined with surgical resection or radiofrequency ablation of liver lesions.

DETAILED DESCRIPTION:
Liver metastases are detected in 40-50% of patients diagnosed with colorectal cancer. Local treatments like surgical resection or radiofrequency ablation result in 5-year survival of 35%. However, relapse still occurs in 70% of patients. Stereotactic body radiotherapy (SBRT) has emerged as a valid treatment not only to provide excellent symptom palliation, but also is effective in local control of metastatic lesions and improves survival. The potential efficacy of SBRT as adjuvant radiotherapy in CRLM patients after surgical resection or radiofrequency ablation is still unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven unresectable metastatic colorectal cancer (CRC)
2. Primary resection of colorectal cancer (CRC)
3. Age≥18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
5. Absence of evidence of extra-hepatic diseases
6. 1 to 3 liver metastases with an individual maximum diameter of up to 5 cm
7. Metastatic liver lesions receiving R0 or R1 resection or radiofrequency ablation with visible tumor bed
8. Aspartate aminotransferase, alanine aminotransferase & alkaline phosphates must be ≤ 2.5 times of the upper limit of normal. Total bilirubin must be within the limit of normal.
9. Patients should have adequate bone marrow function as defined by peripheral granulocyte count of ≥1500/mm3.
10. Patients must provide verbal and written informed consent to participate in the study.
11. Absence of any severe pulmonary or cardiac diseases

Exclusion Criteria:

1. Patients with either untreated brain metastases or brain metastases treated within the past three months are ineligible
2. Patients who are pregnant
3. Patients with severe organ dysfunction
4. History of liver radiotherapy
5. Unwillingness to participate or inability to comply with the protocol for the duration of the study
6. Participation in any investigational drug study within 3 months preceding the start of study treatment
7. Patients not suitable to take part in clinical trials judged by researches

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 2 years
  Evaluate the effect of consolidative SBRT of liver lesions versus observation on disease free survival

SECONDARY OUTCOMES:
Overall survival | 5 years
  To evaluate overall survival after consolidative SBRT in comparison to observation alone
Intrahepatic disease free survival | 2 years
  To evaluate Intrahepatic disease free survival after consolidative SBRT in comparison to observation alone
Toxicities | 2 years
  Acute toxicity was scored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0 criteria during and up to 3 months after radiotherapy. Late toxicity was graded using the Radiation Therapy Oncology Group (RTOG)/European Organisation for the Research and Treatment of Cancer (EORTC) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Nordlinger B, Guiguet M, Vaillant JC, Balladur P, Boudjema K, Bachellier P, Jaeck D. Surgical resection of colorectal carcinoma metastases to the liver. A prognostic scoring system to improve case selection, based on 1568 patients. Association Francaise de Chirurgie. Cancer. 1996 Apr 1;77(7):1254-62. PMID 8608500
- [Result] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196